CLINICAL TRIAL: NCT03854773
Title: Comparison Of Erector Spinae Plane Block And Thoracal Paravertebral Block For Postoperative Analgesia Management Following Vıdeo Assisted Thoracic Surgery
Brief Title: Erector Spinae Plane Block and Thoracal Paravertebral Block Following Video Assisted Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Medical Doctor, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MedipolU
Record Dates: First submitted 2019-02-22; First posted 2019-02-26 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Lung Diseases
Keywords: Erector spinae plane block; Video assisted thoracic surgery,; Postoperative analgesia
MeSH Terms: conditions — Lung Diseases | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: there are three models for this study. the first group is erector spinae plane block group. the second one is thoracal paravertebral block group. the third one is the control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: the patient and the anesthesiologist who performs postoperative pain evaluation will not know the group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Erector spinae block (Group ESPB) (Active Comparator): In group A, ESP block will be performed. US probe will be placed longitudinally 2-3 cm lateral to the T5 transverse process. From superior to inferior, three muscles will be visualized on the hyperechoic transverse process; trapezius (upper), rhomboideus major (middle), erector spinae (lower). The block needle will be inserted cranio caudal direction and then for correction of the needle 5 ml saline will be injected deep into the erector spina muscle fascia. Following confirmation of the correct position of the needle 20 ml %0.25 bupivacaine will be administered for block.
  Interventions: Other: Erector spinae plane block (Group ESPB)
- Thoracal paravertebral block group (Group TPVB) (Active Comparator): In group B, TPVB will be performed. US probe will be placed 2-3 cm laterally following the visualization T5 spinous process in sagittal orientation. The ribs and transverse processes will be visualized as hyperechoic structures. The costotransverse ligament will be visualized in the superior, and the pleura in the anterior region. Using in plane technique, the block needle will be inserted in the cranio-caudal direction until the costotransverse ligament will be passed. For confirmation of correct position of the needle, 5 ml saline will be injected. After the negative aspiration of cerebrospinal fluid, blood and air; 20 ml of 0.25% bupivacaine will be performed and it will be seen of moving downwards of the pleura during the injection
  Interventions: Other: Thoracal paravertebral block (Group TPVB)
- Control group (Group C) (Other): Patients in control group will be only received fentanyl via a patient controlled analgesia (PCA) device.
  Interventions: Other: Control group (group C)

INTERVENTIONS:
Other: Erector spinae plane block (Group ESPB) — Patients will be administered A 400 mg dose of ibuprofen every 8 hours in the postoperative period. A patient controlled device prepared with 10 mcg/ ml fentanyl will be attached to all patients with a protocol included 10 mcg bolus without infusion dose, 10 min lockout time and 4 hour limit. Postoperative patient evaluation will be performed by an anesthesiologist blinded to the procedure.
  Arms: Erector spinae block (Group ESPB)
Other: Thoracal paravertebral block (Group TPVB) — Patients will be administered A 400 mg dose of ibuprofen every 8 hours in the postoperative period. A patient controlled device prepared with 10 mcg/ ml fentanyl will be attached to all patients with a protocol included 10 mcg bolus without infusion dose, 10 min lockout time and 4 hour limit. Postoperative patient evaluation will be performed by an anesthesiologist blinded to the procedure.
  Arms: Thoracal paravertebral block group (Group TPVB)
Other: Control group (group C) — Patients will be administered A 400 mg dose of ibuprofen every 8 hours in the postoperative period. A patient controlled device prepared with 10 mcg/ ml fentanyl will be attached to all patients with a protocol included 10 mcg bolus without infusion dose, 10 min lockout time and 4 hour limit. Postoperative patient evaluation will be performed by an anesthesiologist blinded to the procedure.
  Arms: Control group (Group C)

SUMMARY:
Video assisted thoracic surgery (VATS) has recently been evaluated as the standard surgical procedure for lung surgery. Although VATS is less painful than thoracotomy, patients may feel severe pain during the first hours at postoperative period. Analgesia management is very important for these patients in postoperative period since insufficient analgesia can cause pulmonary complications such as atelectasis, pneumonia and increased oxygen consumption. The ultrasound (US) guided erector spina plane (ESP) block is a novel interfacial plan block defined by Forero et al. at 2016. ESP block provides thoracic analgesia at T5 level and abdominal analgesia at T7-9 level. Visualization of sonoanatomy with US is easy, and the spread of local anesthesic agents can be easily seen under the erector spinae muscle (12). Thus, analgesia occurs in several dermatomes with cephalad-caudad way. In the literature, there is not still any randomized study evaluating ESP block efficiency for postoperative analgesia management after VATS. The aim of this study is to compare US-guided ESP block and TPVB for postoperative analgesia management after VATS.

DETAILED DESCRIPTION:
Video assisted thoracic surgery (VATS) has recently been evaluated as the standard surgical procedure for lung surgery. The advantages of VATS procedures compared with open thoracotomy are rapid recovery, short hospital stay and low complication risk. Although VATS is less painful than thoracotomy, patients may feel severe pain during the first hours at postoperative period. Thoracic epidural analgesia (TEA) which is the gold standard analgesic technique after thoracotomy, is generally used for analgesia management after VATS. However, since the surgical technique and trauma between open surgery and VATS are different, the question of what should be the gold standard for analgesia management after VATS is a topic of discussion. Especially due to the difficult administration and adverse effect profile of TEA, the opinion of minimally invasive surgical procedures, requiring less invasive analgesic techniques is supported. Thoracic paravertebral block (TPVB) has been evaluated as the first step regional analgesia technique for postoperative analgesia management after VATS. However, its administration is difficult because of its anatomical proximity to important structures such as the pleura and central neuro-axial system and it can cause complications such as pneumothorax, vascular injury. Analgesia management is very important for these patients in postoperative period since insufficient analgesia can cause pulmonary complications such as atelectasis, pneumonia and increased oxygen consumption.

The ultrasound (US) guided erector spina plane (ESP) block is a novel interfacial plan block defined by Forero et al. at 2016. ESP block provides thoracic analgesia at T5 level and abdominal analgesia at T7-9 level. The ESP block contains a local anesthetic injection into the deep fascia of erector spinae. This area is away from the pleural and neurological structures and thus minimizes the risk of complications due to injury. Visualization of sonoanatomy with US is easy, and the spread of local anesthesic agents can be easily seen under the erector spinae muscle. Thus, analgesia occurs in several dermatomes with cephalad-caudad way. Cadaveric studies have shown that the injection spreads to the ventral and dorsal roots of the spinal nerves and creates sensory blockade in both posterior and anterolateral thorax. In the literature, it has been reported that ESP block provides effective analgesia after open heart surgery, breast surgery and ventral hernia repair in randomized controlled studies about ESP block efficiency for postoperative analgesia management. In some case series and case reports it has been reported that ESP block provides effective analgesia after thoracotomy and VATS. Furthermore, it has been reported that it provides effective analgesia in chronic and persistant pain syndromes of thorax.

The aim of this study is to compare US-guided ESP block and TPVB for postoperative analgesia management after VATS. The primary aim is to compare perioperative and postoperative opioid consumption and the secondary aim is to evaluate postoperative pain scores (VAS), adverse effects related with opioids (allergic reaction, nausea, vomiting) and complications due to blocks (pneumothorax, hematoma).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II
* scheduled for VATS under general anesthesia

Exclusion Criteria:

* history of bleeding diathesis,
* receiving anticoagulant treatment,
* known local anesthetics and opioid allergy,
* infection of the skin at the site of the needle puncture,
* pregnancy or lactation,
* patients who do not accept the procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
opioid consumption | Change from Baseline Postoperative Visual Analogue Score at 48 hours
  The primary aim is to compare perioperative and postoperative opioid consumption

SECONDARY OUTCOMES:
Visual analogue scores (VAS) | postoperative 1, 2, 4, 8, 16, 24, and 48 hours
  Postoperative pain assessment will be performed using the VAS score (0 = no pain, 10 = the most severe pain felt). The VAS scores at rest and during cough will be recorded at postoperative 1, 2, 4, 8, 16 and 24 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
we will not share IPD

REFERENCES:
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Forero M, Rajarathinam M, Adhikary S, Chin KJ. Continuous Erector Spinae Plane Block for Rescue Analgesia in Thoracotomy After Epidural Failure: A Case Report. A A Case Rep. 2017 May 15;8(10):254-256. doi: 10.1213/XAA.0000000000000478. PMID 28252539
- [Background] Vogt A, Stieger DS, Theurillat C, Curatolo M. Single-injection thoracic paravertebral block for postoperative pain treatment after thoracoscopic surgery. Br J Anaesth. 2005 Dec;95(6):816-21. doi: 10.1093/bja/aei250. Epub 2005 Sep 30. PMID 16199417